CLINICAL TRIAL: NCT05058651
Title: Randomized Phase II/III Trial of First Line Platinum/Etoposide With or Without Atezolizumab (NSC#783608) in Patients With Poorly Differentiated Extrapulmonary Small Cell Neuroendocrine Carcinomas (NEC)
Brief Title: Evaluating the Addition of the Immunotherapy Drug Atezolizumab to Standard Chemotherapy Treatment for Advanced or Metastatic Neuroendocrine Carcinomas That Originate Outside the Lung
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-09851; NCI-2021-09851 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2012 (Other: SWOG); S2012 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2021-09-25; First posted 2021-09-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Advanced Extrapulmonary Neuroendocrine Carcinoma; Metastatic Extrapulmonary Neuroendocrine Carcinoma; Recurrent Extrapulmonary Neuroendocrine Carcinoma; Unresectable Extrapulmonary Neuroendocrine Carcinoma
MeSH Terms: interventions — atezolizumab; Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; Magnetic Resonance Spectroscopy; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm I (atezolizumab, platinum drug, etoposide) (Experimental): During induction phase, patients receive atezolizumab IV over 30-60 minutes on day 1 of each cycle, carboplatin IV over 30 minutes or cisplatin IV over 60 minutes on day 1 of each cycle, and etoposide IV on days 1-3 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. During maintenance phase, patients receive atezolizumab IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI throughout the trial and blood sample collection on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Etoposide; Procedure: Magnetic Resonance Imaging
- Arm II (atezolizumab, platinum drug, etoposide, observation) (Experimental): During induction phase, patients receive atezolizumab IV over 30-60 minutes on day 1 of each cycle, carboplatin IV over 30 minutes or cisplatin IV over 60 minutes on day 1 of each cycle, and etoposide IV on days 1-3 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo observation for 1 year. Patients also undergo CT scan and/or MRI throughout the trial and blood sample collection on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Other: Patient Observation
- Arm III (platinum drug, etoposide, observation) (Active Comparator): During induction phase, patients receive carboplatin IV over 30 minutes or cisplatin IV over 60 minutes on day 1 of each cycle and etoposide IV on days 1-3 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo observation for 1 year. Patients also undergo CT scan and/or MRI throughout the trial and blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Etoposide; Procedure: Magnetic Resonance Imaging; Other: Patient Observation

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
  Arms: Arm I (atezolizumab, platinum drug, etoposide); Arm II (atezolizumab, platinum drug, etoposide, observation)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm II (atezolizumab, platinum drug, etoposide, observation); Arm III (platinum drug, etoposide, observation)

SUMMARY:
This phase II/III trial compares the effect of immunotherapy with atezolizumab in combination with standard chemotherapy with a platinum drug (cisplatin or carboplatin) and etoposide versus standard therapy alone for the treatment of poorly differentiated extrapulmonary (originated outside the lung) neuroendocrine cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). The other aim of this trial is to compare using atezolizumab just at the beginning of treatment versus continuing it beyond the initial treatment. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cisplatin and carboplatin are in a class of medications known as platinum-containing compounds that work by killing, stopping or slowing the growth of cancer cells. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair, and it may kill cancer cells. Giving atezolizumab in combination with a platinum drug (cisplatin or carboplatin) and etoposide may work better in treating patients with poorly differentiated extrapulmonary neuroendocrine cancer compared to standard therapy with a platinum drug (cisplatin or carboplatin) and etoposide alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the combination of induction platinum/etoposide and atezolizumab followed by maintenance atezolizumab (Arm 1) versus induction platinum/etoposide alone (Arm 3).

II. Compare the combination of induction platinum/etoposide and atezolizumab followed by observation (Arm 2) versus induction platinum/etoposide alone (Arm 3).

III. Compare the combination of induction platinum/etoposide and atezolizumab followed by maintenance atezolizumab (Arm 1) versus the combination of induction platinum/etoposide and atezolizumab followed by observation (Arm 2).

SECONDARY OBJECTIVES:

I. To compare overall survival (OS), measured from start of observation/maintenance, across arms.

II. To compare progression free survival (PFS) (measured from randomization and measured from start of observation/maintenance) across arms.

III. To compare objective response rate (ORR = confirmed and unconfirmed partial response [PR] + confirmed and unconfirmed complete response [CR]) across arms among patients with measurable disease at randomization.

IV. To compare clinical benefit rate (CBR = confirmed and unconfirmed PR + confirmed and unconfirmed CR + stable disease [SD]) across arms among patients with measurable disease at randomization.

V. To compare duration of response (DOR) across arms. VI. To evaluate the safety and tolerability of each arm.

ADDITIONAL OBJECTIVE:

I. To bank tumor and blood samples for future biomarker correlative studies.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: During induction phase, patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1 of each cycle, carboplatin IV over 30 minutes or cisplatin IV over 60 minutes on day 1 of each cycle, and etoposide IV on days 1-3 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. During maintenance phase, patients receive atezolizumab IV over 30-60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: During induction phase, patients receive atezolizumab IV over 30-60 minutes on day 1 of each cycle, carboplatin IV over 30 minutes or cisplatin IV over 60 minutes on day 1 of each cycle, and etoposide IV on days 1-3 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo observation for 1 year.

ARM III: During induction phase, patients receive carboplatin IV over 30 minutes or cisplatin IV over 60 minutes on day 1 of each cycle and etoposide IV on days 1-3 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo observation for 1 year.

Patients in all arms also undergo compute tomography (CT) scan and/or magnetic resonance imaging (MRI) throughout the trial and blood sample collection on study.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically-confirmed (local site pathological confirmation sufficient) extrapulmonary poorly differentiated, neuroendocrine carcinoma (NEC)
* Participants must have disease that is unresectable or metastatic and not eligible for definitive therapy as deemed per the treating investigator
* Participants must have radiologically evaluable disease, measurable or non-measurable, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. All measurable and nonmeasurable lesions must be assessed by CT scan with IV contrast of the chest/abdomen/and pelvis (or CT chest without contrast and MRI abdomen/pelvis with gadolinium contrast, if contraindication to CT iodinated contrast) within 28 days prior to registration. While may be used for routine clinical evaluation, PET scans and bone scans alone are not acceptable for disease assessment while participating in this study. All known sites of disease must be assessed and documented on the Baseline Tumor Assessment Form
* Participants must have brain MRI (or CT head with contrast if there is contraindication to MRI brain) if clinically indicated within 28 days prior to registration. Note: Brain imaging is not required in participants without known and/or clinical concern for brain metastases. Participants with asymptomatic central nervous system (CNS) metastases are eligible if one or more of the following apply:

  * Participants who have received treatment for brain metastases must have:

    * No evidence of radiological progression (by MRI brain or CT head with contrast if there is contraindication to MRI brain) within 28 days prior to registration
    * Discontinued all corticosteroids at least 14 days prior to registration
  * Participants with treatment-naive brain lesions must have:

    * No lesion measuring > 2.0 cm in size in any axis
    * MRI brain or CT head with contrast (if there is contraindication to MRI brain) demonstrating no evidence for mass effect, edema, or other impending neurological compromise within 28 days prior to registration
    * No evidence of radiological progression (by MRI brain or CT head with contrast if there is contraindication to MRI brain) within 28 days prior to registration
    * No need for > 2 mg of dexamethasone (or equivalent of > 10 mg prednisone) per day at time of registration
* Participants must not have symptomatic central nervous system (CNS) metastases
* Participants must not have known or suspected leptomeningeal disease
* Participants with prior history of non-metastatic (localized/locally advanced disease) extrapulmonary poorly differentiated NEC may have had prior platinum-based therapy +/- radiation +/- surgery provided that all therapy was completed >= 6 months prior to registration
* Participants must discontinue denosumab prior to study registration and plan to replace with a bisphosphonate while on the study
* Participants must not have had prior treatment for advanced or metastatic NEC EXCEPT one cycle of platinum (carboplatin/cisplatin) + etoposide is allowed prior to registration. Other chemotherapy regimens are not allowed. For participants with prostate or urothelial NEC, prior chemotherapy for the non-NEC component (e.g. adenocarcinoma or urothelial) is allowed as long as such therapy was completed >= 24 weeks prior to registration and participants have recovered from all prior toxicities to =< grade 1.
* Participants must not have had prior treatment with an anti-PD-1, anti-PD-L1, antiPD-L2, CD137 agonists, anti-CTLA-4 agent, or any other immune checkpoint inhibitors for any neuroendocrine neoplasm. Immune checkpoint inhibitors given for other cancer indications are allowed provided last therapy was given at least 12 months prior to study registration
* Participants must not have received treatment with systemic immunostimulatory agents including, but not limited to, interferon and interleukin2 [IL-2] within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to registration
* Participants must not have had history of known severe allergy, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies, including to Chinese hamster ovary cell products or to any component of the atezolizumab formulation, cisplatin, carboplatin, or etoposide
* Participants must not be on active systemic therapy for another cancer with the exception of hormonal therapy including androgen deprivation therapy (e.g., gonadotropin-releasing hormone [GnRH] agonists or antagonists), which can be continued while participants are receiving protocol therapy. Use of enzalutamide or apalutamide is permitted after completion of chemotherapy and must be held during chemotherapy for participants receiving prior to enrollment. Use of darolutamide is permitted during chemotherapy. Glucocorticoid-containing regimens, including abiraterone, are not permitted.
* Participants must be >= 18 years of age
* Participants must have a Zubrod performance status of =< 2 within 28 days prior to registration
* Participants must have a complete medical history and physical exam within 28 days prior to registration
* Absolute neutrophil count (ANC) >= 1.5 x 10^9 /L (obtained within 14 days prior to registration. For participants who received a cycle of chemotherapy prior to registration, at least 21 days must have elapsed between day 1 of platinum + etoposide and performance of these tests)
* Hemoglobin >= 9.0 g/dl (obtained within 14 days prior to registration. For participants who received a cycle of chemotherapy prior to registration, at least 21 days must have elapsed between day 1 of platinum + etoposide and performance of these tests)
* Platelet count >= 100 x 10^9/L (obtained within 14 days prior to registration. For participants who received a cycle of chemotherapy prior to registration, at least 21 days must have elapsed between day 1 of platinum + etoposide and performance of these tests)
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x institutional upper limit of normal (ULN) (obtained within 14 days prior to registration. For participants who received a cycle of chemotherapy prior to registration, at least 21 days must have elapsed between day 1 of platinum + etoposide and performance of these tests)
* Serum total bilirubin =< 1.5 x ULN (obtained within 14 days prior to registration. For participants who received a cycle of chemotherapy prior to registration, at least 21 days must have elapsed between day 1 of platinum + etoposide and performance of these tests)
* Adequate renal function as defined by any 1 of the following: 1) Measured creatinine clearance (CL) > 50 mL/min OR 2) Calculated creatinine CL > 50 mL/min by the Cockcroft-Gault formula OR by 24-hour urine collection for determination of creatinine clearance (obtained within 14 days prior to registration. For participants who received a cycle of chemotherapy prior to registration, at least 21 days must have elapsed between day 1 of platinum + etoposide and performance of these tests)
* Participants must not have uncontrolled or symptomatic hypercalcemia (> 1.5 mmol/L ionized calcium or calcium > 12 mg/dL or corrected serum calcium > ULN) within 14 days prior to registration. Participants who have asymptomatic hypercalcemia are eligible provided that medical therapy to treat the hypercalcemia is planned
* Participants must not have a diagnosis of immunodeficiency nor be receiving systemic steroid therapy (equivalent of > 20 mg of hydrocortisone per day) or any other form of immunosuppressive therapy within 14 days prior to registration
* Participants must not have active or history of autoimmune disease or immune deficiency, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study
  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* Participants must not have history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. NOTE: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Participants must not have significant cardiovascular disease, such as New York Heart Association class II or greater cardiac disease, myocardial infarction within 3 months prior to registration, unstable arrythmias, or unstable angina
* Participants must not have had a major surgical procedure other than for diagnosis within 28 days prior to registration. Participant must not plan to receive a major surgical procedure during the course of protocol treatment. NOTE: Patient port placement is not considered a major surgery
* Participants must not have severe infections (i.e., Common Terminology Criteria for Adverse Events [CTCAE] grade >= 2) at time of registration, including but not limited to hospitalization for complications for infection, bacteremia, or severe pneumonia
* Participants must not have known active tuberculosis
* Participants with evidence of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load, with testing performed as clinically indicated
* Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with active HCV infection who are currently on treatment must have an undetectable HCV viral load, with testing performed as clinically indicated
* Participants with known human immunodeficiency virus (HIV)-infection must be on effective anti-retroviral therapy at time of registration and have undetectable HIV viral load within 6 months of registration
* Participants must not have prior allogeneic bone marrow transplantation or solid organ transplant
* Participants must not have received administration of a live, attenuated vaccine (e.g., FluMist [registered trademark]) within 28 days prior to initiation of study treatment, during treatment with atezolizumab, and not plan to receive for 5 months after the last dose of atezolizumab
* Participants must not be pregnant due to the possibility of harm to the fetus. Individuals who are of reproductive potential must have agreed to use an effective contraceptive method (with details provided as a part of the consent process) during the treatment period and for 5 months after the final dose of atezolizumab. A person who has had menses at any time in the preceding 12 consecutive months or who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a sideeffect of pregnancy prevention) including hysterectomy, bilateral oophorectomy, bilateral tubal ligation/occlusion, and vasectomy with testing showing no sperm in the semen
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of registration or from date of start of observation/maintenance therapy to date of death due to any cause, assessed up to 5 years
  Log-rank tests stratified by the randomization stratification factors will be used for null hypothesis (efficacy) tests. Cox regression models stratified by the randomization stratification factors will be used for alternative hypothesis (futility) tests.

SECONDARY OUTCOMES:
Progression-free survival | From date of registration or start of observation/maintenance therapy to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method and compared using log-rank tests.
Duration of response | Time from date of initial response to date of progression or death, assessed up to 5 years
  Will be estimated non-parametrically using cumulative incidence curves.
Objective response rate (confirmed complete response [CR] or partial response [PR]) | Up to 5 years from study enrollment
  Will be tabulated and compared between arms using Fisher's exact test.
Clinical benefit rate (confirmed CR or PR of any amount of time or stable disease for 6 months or longer) | Up to 5 years from study enrollment
  Will be tabulated and compared between arms using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: David B Zhen, Principal Investigator — SWOG Cancer Research Network
Locations (240):
- United States (240):
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente-Ontario, Ontario, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Woodland Memorial Hospital, Woodland, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - AdventHealth Porter, Denver, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Levine Cancer Institute-SouthPark, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm